CLINICAL TRIAL: NCT06656559
Title: Endoscopic Retrograde Cholangiopancreatography With Radiofrequency Ablation (ERCP-RFA) Combined With Envafolimab and Surufatinib Sequential Therapy for Unresectable Biliary Tract Carcinoma: A Prospective, Single-Arm, Single-Center Phase II Clinical Study
Brief Title: Endoscopic Retrograde Cholangiopancreatography With Radiofrequency Ablation (ERCP-RFA) Combined With Envafolimab and Surufatinib Sequential Therapy for Unresectable Biliary Tract Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2024-0131
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Unresectable Biliary Tract Carcinoma
MeSH Terms: interventions — envafolimab; surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab and Surufatinib (Experimental)
  Interventions: Drug: Envafolimab and Surufatinib

INTERVENTIONS:
Drug: Envafolimab and Surufatinib — Envafolimab: 150mg, SC, qw Surufatinib: 150mg, p.o., qd

SUMMARY:
The sequential treatment strategy of ERCP-RFA combined with envafolimab and surufatinib proposed in this study aims to maximally inhibit the progression of unresectable biliary tract tumors through the combined application of multiple therapeutic modalities. ERCP-RFA, as a local treatment, first reduces the tumor burden and alleviates biliary obstruction through physical ablation. Subsequently, Envafolimab enables the body to more effectively identify and attack the remaining tumor cells by activating the immune system. Finally, Surufatinib as a targeted drug, further controls the growth and spread of tumors by inhibiting tumor angiogenesis and cell proliferation. The potential advantage of this combined treatment lies in the complementary effects of different therapeutic modalities.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent.;
* 18-79 years of age (at the time of signing the informed consent);
* Patients with confirmed diagnosis of biliary tract tumors by histopathologic examination;
* Patients have received no previous local treatment or any systemic treatment, and have been considered unsuitable for radical therapies
* Patients assessed by the investigator as unsuitable for or refusing chemotherapy
* At least one measurable lesion (≥10 mm long diameter on CT scan for tumor lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to RECIST 1.1 criteria);
* ECOG score: 0-1;
* Expected survival ≥ 12 weeks;
* Vital organ function in accordance with the following requirements (excluding any blood components and cell growth factors within 14 days): 1) blood routine: neutrophils ≥ 1.5 × 10^9/L platelet count ≥ 60 × 10^9/L hemoglobin ≥ 90 g/L; 2) liver and kidney function: serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); total bilirubin (TBIL) ≤ 1.5 times ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 ULN (≤ 5ULN if liver function abnormalities are due to liver metastases); urine protein < 2 +; if urine protein ≥ 2 +,24-hour urine protein must show protein ≤ 1g;
* Normal coagulation, no active bleeding and thrombosis disease 1) international normalized ratio INR ≤ 1.5 × ULN; 2) partial thromboplastin time APTT ≤ 1.5 × ULN; 3) prothrombin time PT ≤ 1.5 × ULN;
* Non-surgically sterilized or female patients of childbearing age who need to use a medically recognized contraceptive (such as an intrauterine device, contraceptive pills or condom) during study treatment and within 3 months after the end of study treatment; non-surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 7 days before study enrollment; and must be non-lactating; non-surgically sterilized or male patients of childbearing age who need to agree to use a medically recognized contraceptive during study treatment and within 3 months after the end of study treatment with their spouses.
* Willing and able to be followed up until death or end of study or study termination.

Exclusion Criteria:

* History of other malignancies (except basal cell carcinoma of the skin and/or carcinoma in situ of the cervix after radical surgery).
* Previous treatment with other immune checkpoints; the subject known to have a prior allergy to macromolecular protein preparations;
* Presence of any active autoimmune disease or history of autoimmune disease in the subject;
* Subjects who are on immunosuppressive, or systemic, or absorbable topical hormone therapy for immunosuppression (dose >10mg/day prednisone or other equipotent hormone) and who continue to be on it within 2 weeks prior to enrollment.
* Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites that require repeated drainage;
* Patients with poorly controlled cardiac clinical symptoms or diseases such as: (1) NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* Subjects with active infection or unexplained fever >38.5 degrees Celsius during screening and prior to the first dose (if the subject had fever due to the tumor, as determined by the investigator, he could be enrolled);
* Previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc.;
* Subjects with congenital or acquired immune deficiency (e.g., HIV-infected individuals)
* Subjects who have had a live bacterial vaccine or live attenuated vaccine vaccine within 4 weeks prior to the first dose of study treatment.
* Subject has a known history of psychiatric drug abuse, alcoholism, or drug abuse;
* Patients who cannot be administered orally
* The subject had received treatment with traditional Chinese medicine within 2 weeks before the first treatment
* ECOG score: ≥2
* Patients with any other diseases, dysfunction caused by metastatic lesions, or suspected disease found by physical examination, indicating possible contraindications to the use of the investigational drug or putting the patients at high risk of treatment-related complications.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | up to 12 months
  Defined as the time from the start of study treatment to death due to any cause

SECONDARY OUTCOMES:
Disease Control Rate | up to 12 months
  Complete response(CR)and partial response(PR)
Progression-Free Survival | up to 12 months
  Assessed by the investigator using RECIST v1.1, defined as the time from the start of study treatment to disease progression, or relapse after resection of liver metastases, or death due to any cause.
Overall Response Rate | up to 12 months
  Partial response (PR) plus complete response (CR)): assessed by the investigator using RECIST v1.1 criteria
Adverse events was evaluated during received protocol therapy according to the NCI Common Terminology Criteria for NCI- CTCAE 5.0. | up to 12 months
  safety

IPD SHARING:
Plan to Share IPD: No